CLINICAL TRIAL: NCT02849509
Title: Non-interventional Study Describing Patients' Perception on Anticoagulant Treatment and Treatment Convenience When Treated With Pradaxa or Vitamin K Antagonist for Stroke Prophylaxis in Atrial Fibrillation.
Brief Title: Patient Convenience Study- NIS RELATE
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.261
Record Dates: First submitted 2016-05-04; First posted 2016-07-29 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Switch Patients / A: Patients with non-valvular atrial fibrillation (NVAF), currently on Vitamin K Antagonist (VKA) therapy, who are switched to Pradaxa.
  Interventions: Drug: Pradaxa (dabigatran)
- New Patients / B: Newly diagnosed NVAF patients who are treated with VKA or Pradaxa (VKA : Pradaxa = 1:1).
  Interventions: Drug: Vitamin K antagonist

INTERVENTIONS:
Drug: Pradaxa (dabigatran) — Pradaxa (dabigatran etexilate)110mg or 150mg
  Groups: Switch Patients / A
Drug: Vitamin K antagonist — Vitamin K antagonist or Pradaxa
  Groups: New Patients / B

SUMMARY:
The aim of this non-interventional study is to describe patient's perception of anticoagulant treatment when using Pradaxa® to prevent stroke and systemic embolism while suffering from atrial fibrillation (according to its approved indication in the approved dosages of 110 mg or 150 mg twice daily) in comparison to standard care using Vitamin K Antagonist (VKA).

ELIGIBILITY:
Inclusion criteria:

Cohort A:

1. A. Written informed consent prior to participation
2. A. Female and male patients >= 18 years of age with a diagnosis of non-valvular atrial fibrillation.
3. A. At least 3 months of continuous VKA treatment for stroke prevention prior to baseline assessment.
4. A. Patients switched to Pradaxa® according Summary of Product Characteristics and physician's discretion.

OR

Cohort B:

1. B. Written informed consent prior to participation.
2. B. Female and male patients >= 18 years of age newly diagnosed with non-valvular atrial fibrillation and no previous treatment for stroke prevention (no use of any oral anticoagulant (OAC) within one year prior to enrolment).
3. B. Stroke prevention treatment initiated with Pradaxa® or VKA according to Summary of Product Characteristics and physician's discretion.

Exclusion criteria:

1. Contraindication to the use of Pradaxa® or VKA as described in the Summary of Product Characteristics (SmPC).
2. Patients receiving Pradaxa® or VKA for any other condition than stroke prevention in atrial fibrillation.
3. Current participation in any clinical trial of a drug or device.
4. Current participation in an European registry on the use of oral anticoagulation in AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SEASK Patients with Non valvuar Atrial Fribrillation
Sampling Method: Non-Probability Sample
Enrollment: 1313 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (50):
- Indonesia (3):
  - Harapan Kita National Cardiovascular Center, Jakarta Barat
  - Rumah Sakit Bina Waluya, Jakarta Timur
  - Rumah Sakit Siloam Lippo Karawaci, Tangerang, Tangerang
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star
  - Institut Jantung Negara, Kuala Lumpur
  - Hospital University Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - UiTM Sg Buloh Campus, Sg Buloh
- Singapore (2):
  - National Heart Center, Singapore
  - Changi General Hospital, Singapore
- South Korea (33):
  - Korea University Ansan Hospital, Ansan
  - Sejong General Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National Univ. Hosp, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Dankook University Hospital, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National Univ. Hosp, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejoen
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Wonkwang University School of Medicine & Hospital, Iksan
  - Inha University Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - VHS Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hosp, Wŏnju
- Thailand (6):
  - Bhumibol Adulyadej Hospital, Bangkok
  - King Chulalongkorn Hospital, Bangkok
  - Pramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Chiangmai University, Chiang Mai
  - Thammasat University Hospital, Pathum Tani

REFERENCES:
- [Derived] Lee YS, Oh YS, Choi EK, Chern AKC, Jiampo P, Chutinet A, Hanafy DA, Trivedi P, Zhai D. Patient perception and treatment convenience of dabigatran versus vitamin K antagonist when used for stroke prophylaxis in atrial fibrillation: Real-world Evaluation of Long-term Anticoagulant Treatment Experience (RE-LATE) study. Open Heart. 2021 Dec;8(2):e001745. doi: 10.1136/openhrt-2021-001745. PMID 34857666

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Switch Patients - Pradaxa): Patients with non-valvular atrial fibrillation (NVAF), who were treated with a Vitamin K Antagonist (VKA) therapy for at least 3 months for stroke prevention and then switched to 110 or 150 milligram (mg) twice daily dose of Pradaxa.
- Cohort B (New Patients - Pradaxa): Newly diagnosed NVAF patients who were not previously treated with an anticoagulant for the prevention of stroke, and were initiated on 110 or 150 mg twice daily Pradaxa
- Cohort B (New Patients - VKA): Newly diagnosed NVAF patients who were not previously treated with an anticoagulant for the prevention of stroke, and were initiated on VKA therapy. The choice of vitamin K antagonist and the appropriate dosing was at the discretion of the physician.
Period: Overall Study
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Started | 379 | 591 | 343
Completed | 289 (Not prematurely discontinued from Pradaxa or VKA) | 425 (Not prematurely discontinued from Pradaxa or VKA) | 258 (Not prematurely discontinued from Pradaxa or VKA)
Not Completed | 90 | 166 | 85
Not completed — Worsening of disease under study | 1 | 1 | 1
Not completed — Worsening of other pre-existing disease | 0 | 1 | 2
Not completed — Other adverse event | 36 | 41 | 8
Not completed — Withdrawal by Subject | 6 | 17 | 12
Not completed — Lost to Follow-up | 27 | 67 | 36
Not completed — Other, reason not specified | 14 | 29 | 25
Not completed — No inform. on termination of Pradaxa/VKA | 6 | 10 | 1

BASELINE CHARACTERISTICS:
Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA) | Total
Number analyzed (Participants) | 379 | 591 | 343 | 1313
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Years | 69.7 (9.0) | 67.3 (9.8) | 63.4 (10.9) | 67.0 (10.2)
Age, Customized [Count of Participants; unit: Participants] — Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries
  Participants
    < 65 Years | 95 | 196 | 184 | 475
    >= 65 and < 75 Year | 154 | 256 | 101 | 511
    >= 75 Years | 130 | 139 | 58 | 327
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Female | 130 | 228 | 106 | 464
    Male | 249 | 363 | 237 | 849
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Non-South Korea includes four countries, and they are Indonesia, Malaysia, Singapore, and Thailand. Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries
  Participants
    Korea, Republic Of: Non-South Korea | 54 | 124 | 32 | 210
    Korea, Republic Of: South Korea | 325 | 467 | 311 | 1103
Type of hospital or practice [Count of Participants; unit: Participants] — Type of hospital or practice (Healthcare system characteristics) Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Public | 171 | 255 | 133 | 559
    Private | 200 | 309 | 201 | 710
    Other | 8 | 27 | 9 | 44
Owner of medical practice [Count of Participants; unit: Participants] — Owner of medical practice (Healthcare system characteristics) Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Physician or physician group | 174 | 268 | 162 | 604
    Health Maintenance Organisation (HMO) | 0 | 0 | 0 | 0
    Community health center | 3 | 5 | 2 | 10
    Medical / academic health center | 156 | 231 | 144 | 531
    Other hospital | 22 | 43 | 35 | 100
    Other health care corporation | 0 | 0 | 0 | 0
    Other | 24 | 44 | 0 | 68
Speciality of treating physician [Count of Participants; unit: Participants] — Speciality of treating physician (Healthcare system characteristics) Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Cardiologist | 362 | 572 | 323 | 1257
    General practitioner | 0 | 3 | 1 | 4
    Other specialist | 17 | 16 | 19 | 52
Baseline creatinine clearance category [Count of Participants; unit: Participants] — Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries
  Participants
    <30 mL/min | 0 | 0 | 13 | 13
    30 to <50 mL/min | 64 | 66 | 29 | 159
    50 to <80 mL/min | 126 | 210 | 78 | 414
    >=80 mL/min | 69 | 140 | 69 | 278
    Missing | 120 | 175 | 154 | 449
CHA2DS2-VASc score [Count of Participants; unit: Participants] — CHA2DS2-VASc score: Congestive heart failure, Hypertension, Age (≥ 75), Diabetes mellitus, Stroke/Transient Ischaemic Attack (TIA), Vascular disease, Age 65-74, Sex category. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome. Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Low risk (score=0) | 5 | 29 | 50 | 84
    Intermediate risk (score=1) | 43 | 78 | 106 | 227
    High risk (score ≥2) | 331 | 482 | 187 | 1000
    Missing | 0 | 2 | 0 | 2
HAS-BLED score [Count of Participants; unit: Participants] — HAS-BLED score: Hypertension, Abnormal renal and liver function, Stroke, Bleeding history or predisposition, Labile International Normalized Ratio (INR), Elderly (>65 years), Drugs and Alcohol. HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome. Population: The population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
  Participants
    Low risk (score <3) | 291 | 540 | 306 | 1137
    High risk (score ≥3) | 88 | 49 | 37 | 174
    Missing | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Perception of Anticoagulant Treatment Questionnaire, Part 2 (PACT-Q2) Scores, for Patients in Cohort A, at Second Assessment Compared to Baseline Assessment
Description: Mean Perception of Anticoagulant treatment Questionnaire, part 2 (PACT-Q2) scores, for patients in cohort A, at second assessment compared to baseline assessment. The PACT-Q2 is composed of 3 dimensions covering: convenience (11 items), burden of disease & treatment (2 items), & anticoagulant treatment satisfaction (7 items). In this outcome the mean convenience & satisfaction dimension scores of PACT-Q2 at second assessment (Visit 2) were compared with baseline assessment (Visit 1). Within the PACT-Q2, items for convenience & for burden of disease and treatment were reversed (reversed score = 6 - item score), added together & rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction were summed & rescaled on 0-100 scale to determine satisfaction score. High scores are more favorable.
  PACT-Q2 which were completed more than 1 day after discontinuation of treatment or using incorrect procedure were excluded from analysis.
Time Frame: Visit 1 (Baseline) and second assessment Visit 2 (7-124 days after initiation on Pradaxa or VKA)
Population: The main analysis population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort A (Switch Patients - Pradaxa)
Number analyzed (Participants) | 379
Unit on scale
  Convenience dimension score: Baseline: number analyzed (Participants) | 377
  Convenience dimension score: Baseline | 71.4 (21.8)
  Convenience dimension score: Second assessment: number analyzed (Participants) | 317
  Convenience dimension score: Second assessment | 79.6 (18.1)
  Satisfaction dimension score: Baseline: number analyzed (Participants) | 377
  Satisfaction dimension score: Baseline | 61.0 (13.3)
  Satisfaction dimension score: Second assessment: number analyzed (Participants) | 317
  Satisfaction dimension score: Second assessment | 63.2 (14.6)
Statistical Analysis 1: Comparison: Cohort A (Switch Patients - Pradaxa); Convenience dimension score of PACT-Q2 at the second assessment (Visit 2) were compared with the baseline assessment (Visit 1). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p < 0.0001, Paired t-test — p-value of paired t-test compared to baseline
Statistical Analysis 2: Comparison: Cohort A (Switch Patients - Pradaxa); Satisfaction dimension score of PACT-Q2 at the second assessment (Visit 2) were compared with the baseline assessment (Visit 1). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.0174, Paired t-test — p-value of paired t-test compared to baseline

2. Primary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort A, at Last Assessment Compared to Baseline Assessment
Description: Mean PACT-Q2 scores, for patients in cohort A, at last assessment compared to baseline assessment. The mean convenience and satisfaction dimension scores of PACT-Q2 at the last assessment (Visit 3) were compared with the baseline assessment (Visit 1). Within the PACT-Q2, items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction were summed and rescaled on a 0-100 scale to determine the satisfaction score. High scores are more favorable.
  PACT-Q2 which were completed more than 1 day after discontinuation of treatment or using incorrect procedure were excluded from the analysis.
Time Frame: Visit 1 (Baseline) and last assessment Visit 3 (125-365 days after initiation on Pradaxa or VKA)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort A (Switch Patients - Pradaxa)
Number analyzed (Participants) | 379
Unit on scale
  Convenience dimension score: Baseline: number analyzed (Participants) | 377
  Convenience dimension score: Baseline | 71.4 (21.8)
  Convenience dimension score: Last assessment: number analyzed (Participants) | 266
  Convenience dimension score: Last assessment | 82.0 (16.8)
  Satisfaction dimension score: Baseline: number analyzed (Participants) | 377
  Satisfaction dimension score: Baseline | 61.0 (13.3)
  Satisfaction dimension score: Last assessment: number analyzed (Participants) | 266
  Satisfaction dimension score: Last assessment | 64.4 (14.7)
Statistical Analysis 1: Comparison: Cohort A (Switch Patients - Pradaxa); Convenience dimension score of PACT-Q2 at the last assessment (Visit 3) were compared with the baseline assessment (Visit 1). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p < 0.0001, Paired t-test — p-value of paired t-test compared to baseline
Statistical Analysis 2: Comparison: Cohort A (Switch Patients - Pradaxa); Satisfaction dimension score of PACT-Q2 at the last assessment (Visit 3) were compared with the baseline assessment (Visit 1). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.0004, Paired t-test — p-value of paired t-test compared to baseline

3. Primary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort B, at Second Assessment Compared Between Treatment Groups
Description: Mean PACT-Q2 scores, for patients in cohort B, at second assessment compared between treatment groups. Convenience dimension score and satisfaction dimension score of PACT-Q2 both range from 0 to 100 with high scores indicate better outcome.
  Mean PACT-Q2 scores, for patients in Cohort B, were compared between matched Pradaxa® and VKA patients at the second assessment. The mean convenience and satisfaction scores of PACT-Q2 were compared between matched Pradaxa® and VKA patients. Pradaxa® and VKA patients were matched based on propensity scores using a variable ratio, parallel, balanced 2:1, nearest neighbour matching algorithm with a caliper width of 0.05 and without replacement.
  PACT-Q2 which were completed more than 1 day after discontinuation of treatment or using incorrect procedure were excluded from the analysis.
Time Frame: Second assessment Visit 2 (7-124 days after initiation on Pradaxa or VKA)
Population: The main analysis population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries and propensity score matched patients.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 591 | 343
Unit on scale
  Convenience dimension score: number analyzed (Participants) | 217 | 217
  Convenience dimension score | 78.4 (14.6) | 75.1 (19.6)
  Satisfaction dimension score: number analyzed (Participants) | 217 | 217
  Satisfaction dimension score | 61.5 (12.7) | 59.9 (13.5)
Statistical Analysis 1: Comparison: Cohort B (New Patients - Pradaxa) vs Cohort B (New Patients - VKA); Convenience dimension score of PACT-Q2 for patients in Cohort B, were compared between matched Pradaxa® and VKA patients at the second assessment. There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.0423, Paired t-test — p-value of paired t-test compared between matched Pradaxa® and VKA patients
Statistical Analysis 2: Comparison: Cohort B (New Patients - Pradaxa) vs Cohort B (New Patients - VKA); Satisfaction dimension score of PACT-Q2 for patients in Cohort B, were compared between matched Pradaxa® and VKA patients at the second assessment. There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.2226, Paired t-test — p-value of paired t-test compared between matched Pradaxa® and VKA patients

4. Primary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort B, at Last Assessment Compared Between Treatment Groups
Description: Mean PACT-Q2 scores, for patients in cohort B, at last assessment compared between treatment groups.
  Convenience dimension score and satisfaction dimension score of PACT-Q2 both range from 0 to 100 with high scores indicate better outcome.
  Mean PACT-Q2 scores, for patients in Cohort B, were compared between matched Pradaxa® and VKA patients at the last assessment. The mean convenience and satisfaction scores of PACT-Q2 were compared between matched Pradaxa® and VKA patients. Pradaxa® and VKA patients were matched based on propensity scores using a variable ratio, parallel, balanced 2:1, nearest neighbour matching algorithm with a caliper width of 0.05 and without replacement.
Time Frame: Last assessment - Visit 3 (125-365 days after initiation on Pradaxa or VKA)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 591 | 343
Unit on scale
  Convenience dimension score: number analyzed (Participants) | 157 | 157
  Convenience dimension score | 80.4 (13.6) | 76.0 (18.9)
  Satisfaction dimension score: number analyzed (Participants) | 157 | 157
  Satisfaction dimension score | 63.9 (11.6) | 60.9 (12.8)
Statistical Analysis 1: Comparison: Cohort B (New Patients - Pradaxa) vs Cohort B (New Patients - VKA); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0287, Paired t-test — p-value of paired t-test compared between matched Pradaxa® and VKA patients
Statistical Analysis 2: Comparison: Cohort B (New Patients - Pradaxa) vs Cohort B (New Patients - VKA); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.0300, Paired t-test — p-value of paired t-test compared between matched Pradaxa® and VKA patients

5. Primary Outcome: Patient Characterization at Baseline - Categorical Parameters
Description: Categorical parameters of the patient characteristics at baseline included age, gender, Stroke- and/or bleeding related risk factors in medical history (MH), co-morbidities (CoMo), concomitant therapies (CM) and dosing of Pradaxa® (DoP).
Time Frame: Baseline (Visit1)
Population: Eligible patients who took the prescribed treatment and without an important protocol violation
Measure: Number; unit: Percentage of participant
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 379 | 591 | 343
Percentage of participant
  < 65 Years | 25.1 | 33.2 | 53.6
  >= 65 and < 75 Years | 40.6 | 43.3 | 29.4
  >= 75 Years | 34.3 | 23.5 | 16.9
  Female | 34.3 | 38.6 | 30.9
  Male | 65.7 | 61.4 | 69.1
  MH: Thromboembolism | 6.3 | 3.4 | 1.5
  MH: Cardiovascular Conditions | 7.7 | 5.1 | 4.4
  MH: Bleedings | 2.6 | 1.0 | 0.9
  MH: Other Conditions | 5.8 | 3.7 | 3.8
  CoMo: Thromboembolism | 9.8 | 4.7 | 7.6
  CoMo: Cardiovascular Conditions | 64.1 | 50.9 | 40.5
  CoMo: Bleedings | 2.4 | 2.5 | 2.3
  CoMo: Other Conditions | 26.9 | 20.8 | 17.8
  CM:Antihypertensives | 67.5 | 56.0 | 47.8
  CM:Lipid modifying agents | 46.7 | 33.5 | 28.0
  CM:Antithrombotic agents | 15.3 | 9.5 | 19.8
  CM:Proton pump inhibitors | 16.4 | 13.9 | 7.9
  CM:Amiodarone | 7.4 | 7.1 | 5.8
  CM:H2-receptor antagonists | 8.7 | 7.1 | 2.0
  CM:NSAIDS | 1.8 | 2.9 | 1.7
  CM:Verapamil | 1.1 | 1.5 | 1.7
  DoP:110 mg twice daily: number analyzed (Participants) | 379 | 591 | 0
  DoP:110 mg twice daily | 68.1 | 58.0 |
  DoP:150 mg twice daily: number analyzed (Participants) | 379 | 591 | 0
  DoP:150 mg twice daily | 31.9 | 42.0 |

6. Secondary Outcome: Patient Characteristics at Baseline - CHA2DS2-VASc Stroke Risk Score
Description: CHA2DS2-VASc stroke risk score is calculated based on the following conditions: Congestive heart failure, Hypertension, Age (≥ 75), Diabetes Mellitus, Stroke/ Transient Ischaemic Attack (TIA), Vascular disease, Age 65-74, Sex category.
  CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: Baseline (Visit1)
Population: Eligible patients who took the prescribed treatment and without an important protocol violation
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 379 | 589 | 343
unit on scale | 3.1 (1.4) | 2.6 (1.4) | 2.0 (1.6)

7. Secondary Outcome: Patient Characteristics at Baseline - HAS-BLED Bleeding Risk Score
Description: HAS-BLED bleeding risk score is calculated based on the following conditions: Hypertension, Abnormal renal and Hypertension, Abnormal renal and liver function, Stroke, Bleeding history or predisposition, Labile INR, Elderly (>65 years), Drugs and Alcohol.
  HAS-BLED bleeding risk score may range from 0 to 9 with 0 being the best outcome.
Time Frame: Baseline (Visit1)
Population: Eligible patients who took the prescribed treatment and without an important protocol violation
Measure: Mean (Standard Deviation); unit: unit on scale
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 379 | 589 | 343
unit on scale | 1.8 (1.1) | 1.3 (0.9) | 1.1 (1.1)

8. Secondary Outcome: Patient Characteristics at Baseline - Creatinine Clearance
Description: Creatinine clearance at baseline is a measure of the patient's kidney function and is one of the baseline patient characteristics.
Time Frame: Baseline (Visit1)
Population: Eligible patients who took the prescribed treatment and without an important protocol violation
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 259 | 416 | 189
mL/min | 68.114 (23.147) | 75.367 (29.028) | 73.017 (29.179)

9. Primary Outcome: Patient Characteristics at Baseline - Duration of Previous VKA Treatment for Cohort A
Description: Duration of continuous VKA treatment for stroke prevention prior to baseline assessment (Cohort A)
Time Frame: Baseline (Visit1)
Population: Eligible patients who took the prescribed treatment and without an important protocol violation
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Cohort A (Switch Patients - Pradaxa)
Number analyzed (Participants) | 379
Years | 4.28 (3.63)

10. Secondary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort A, at Last Assessment Compared to Second Assessment
Description: Mean PACT-Q2 scores, for patients in cohort A, at last assessment compared to second assessment.
  The PACT-Q2 is composed of 3 dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items).
  The mean convenience and satisfaction dimension scores of PACT-Q2 at the last assessment (Visit 3)were compared with the second assessment (Visit 2). Within the PACT-Q2, items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction were summed and rescaled on a 0-100 scale to determine the satisfaction score.
Time Frame: Second assessment - Visit 2 (7-124 days after initiation on Pradaxa or VKA) and last assessment - Visit 3 (125-365 days after initiation on Pradaxa or VKA)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort A (Switch Patients - Pradaxa)
Number analyzed (Participants) | 379
Unit on scale
  Convenience dimension score (Visit 2) | 79.6 (18.1)
  Convenience dimension score (Visit 3) | 82.0 (16.8)
  Satisfaction dimension score (Visit 2) | 63.2 (14.6)
  Satisfaction dimension score (Visit 3) | 64.4 (14.7)
Statistical Analysis 1: Comparison: Cohort A (Switch Patients - Pradaxa); Convenience dimension score of PACT-Q2 for patients in Cohort A, were compared between second assessment (Visit 2) and last assessment (Visit 3). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.1234, Paired t-test — p-value of paired t-test compared between second assessment (Visit 2) and last assessment (Visit 3)
Statistical Analysis 2: Comparison: Cohort A (Switch Patients - Pradaxa); Satisfaction dimension score of PACT-Q2 for patients in Cohort A, were compared between second assessment (Visit 2) and last assessment (Visit 3). There was no (confirmatory) hypothesis testing foreseen in a strict statistical sense. Analyses were descriptive in nature and p-values from statistical models were used for exploratory purposes; Test type: Other; p = 0.9740, Paired t-test — p-value of paired t-test compared between second assessment (Visit 2) and last assessment (Visit 3)

11. Secondary Outcome: Description of Perception of Anticoagulant Treatment Questionnaire, Part 1 (PACT-Q1) Items at Baseline for Cohort B
Description: For Cohort B, scores of PACT-Q1 at baseline were summarised descriptively.
  The PACT-Q1 is composed of a single dimension (7 items) covering the expectations of patients regarding their anticoagulant treatment and is to be administered before treatment initiation.
  The PACT-Q1 scores ranged from 1 (Not at all) to 5 (Extremely/Completely/ Very much).
Time Frame: Baseline (Visit1)
Population: The main analysis population consisted of all eligible patients (that is, all patients who took the prescribed treatment and without an important protocol violation) from all participating countries. PACT-Q1 data which were collected after the first dose or using incorrect procedure were excluded from the summary.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
Number analyzed (Participants) | 580 | 340
Unit on scale
  A1 - Confidence in prevention of blood clots | 3.4 (1.0) | 3.3 (1.0)
  A2 - Expectations of symptom relief | 3.4 (0.9) | 3.3 (1.0)
  A3 - Expectations of side effects | 2.5 (1.0) | 2.6 (1.0)
  A4 - Importance of ease of use | 3.7 (0.9) | 3.5 (1.0)
  A5 - Worries about making mistakes | 2.5 (1.2) | 2.5 (1.2)
  A6 - Importance of independency | 3.7 (0.9) | 3.7 (1.0)
  A7 - Worries about cost | 2.7 (1.2) | 2.6 (1.2)

ADVERSE EVENTS:
Time Frame: From the first administration of study medication until end of the study, up to 406 days
Description: In this non-interventional study, a systematic collection of safety data was neither planned nor performed. The focus was on non-serious and serious adverse drug reactions to Pradaxa® and VKA and on fatal adverse events (AEs), that is, AEs that were not considered to have a reasonable possibility to be causally related to the prescribed anticoagulant treatment were only collected when fatal
Arm/Group | Cohort A (Switch Patients - Pradaxa) | Cohort B (New Patients - Pradaxa) | Cohort B (New Patients - VKA)
All-Cause Mortality (participants affected / at risk) | 1/379 | 0/591 | 0/343
Serious Adverse Events (participants affected / at risk) | 5/379 | 1/591 | 6/343
Other Adverse Events (participants affected / at risk) | 0/379 | 0/591 | 0/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Switch Patients - Pradaxa) (N=379) | Cohort B (New Patients - Pradaxa) (N=591) | Cohort B (New Patients - VKA) (N=343)
International normalised ratio increased (Investigations) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The choice of anticoagulant treatment was at the discretion of the treating physician and independent from study participation. The planned between-country comparisons of study results could not be performed or were not meaningful when performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02849509/SAP_000.pdf
  • Study Protocol (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT02849509/Prot_001.pdf